CLINICAL TRIAL: NCT01676558
Title: A Phase II Study of 131I-rituximab for Elderly or Poor Performance Status Patients With Diffuse Large B Cell Lymphoma (DLBCL) or for Adult Patients With Relapsed or Refractory DLBCL
Brief Title: A Phase II Study of 131I-rituximab for Relapsed/Refractory Diffuse Large B Cell Lymphoma (DLBCL)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Korea Cancer Center Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DLBCL_131I-rituximab RIT
Record Dates: First submitted 2012-08-24; First posted 2012-08-31 (Estimated); Last update posted 2012-11-14 (Estimated); Status verified 2012-08

CONDITIONS: Relapsed or Refractory Diffuse Large B Cell Lymphoma
Keywords: diffuse large B cell lymphoma; radioimmunotherapy; 131I-rituximab
MeSH Terms: conditions — Recurrence; Lymphoma, Large B-Cell, Diffuse | interventions — 131I-rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 131I-rituximab (Experimental): 131I-rituximab treatment interval at least 4 weeks up to maximum 6 cycles
  Interventions: Drug: 131I-rituximab

INTERVENTIONS:
Drug: 131I-rituximab

SUMMARY:
Diffuse large B cell lymphoma (DLBCL) is the most common type of non-Hodgkin lymphoma in Korea. Although there is standard therapy, which is called 'R-CHOP', many obstacles to use aggressive cytotoxic chemotherapeutic agents such as old age, poor performance status, refractoriness, and relapsed disease still remains. So we investigate the efficacy of radioimmunotherapy using 131I-rituximab in refractory or relapsed patients with DLBCL.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diffuse large B cell lymphoma Elderly (>65 years) or medically ineligible to standard cytotoxic chemotherapy due to poor performance status, or relapsed or refractory patients Eastern Cooperative Oncology Group performance status ≤ 2, age≥ 20 years Relapsed or refractory after autologous hematopoietic stem cell transplantation (auto-HSCT) in young patients with good performance status and indicated to high dose chemotherapy and auto-HSCT More than one measurable lesion
* More than 2cm sized lesion in conventional CT scan,
* More than 1cm sized lesion in spiral CT or contrast-enhanced PET/CT Adequate renal function (serum creatinine ≤ 2.0 mg/dl or Ccr ≥ 60 ml/min) Adequate hepatic function (serum bilirubin ≤ 2.0 mg/dl , AST/ALT ≤ 3 upper normal limit) Adequate bone marrow reservoir (ANC ≥1,500/㎕, platelet count≥ 75,000/㎕) patient who agree the purpose and intention of this clinical trial

Exclusion Criteria:

* recent (<5 years) history of other malignancy or unrecovered from the disease (appropriately treated skin cancer and uterine cervix carcinoma in situ are excluded)

  * hemodynamically unstable due to the recent (<12 months) history of severe heart disease such as myocardial infarction
  * acute complications of severe lung or metabolic disease
  * Combined severe neurological or psychiatric disease Unrecovered from infection or other medical disease Recent (<30 days) history of enrollment of other clinical trial Pregnant or breast-feeding woman women of childbearing potential and men not employing adequate contraception at least for 1 year Previous history drug allergy to the content of 131I-rituximab Infection(sepsis, pneumonia, viral infection, etc) (inactivated hepatitis B carrier can be enrolled) Young patient with good performance status indicated to autologous hematopoietic stem cell transplantation irrespective of the failure of 1st line chemotherapy

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2012-06; Primary Completion 2016-06 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
overall response rate | up to 5 years
  International Working Group Response criteria

SECONDARY OUTCOMES:
Response duration | up to 5 years
progression free survival | up to 5 years
Overall survival | up to 5 years
Number of Adverse event | up to 5 years
  grading the adverse events using CTCAE version 4.03

CONTACTS AND LOCATIONS:
Locations (1):
- Korea Cancer Center Hospital, Korea Institute of Radiological and Medical Sciences, Seoul, South Korea